CLINICAL TRIAL: NCT05615779
Title: The Fibre Study: RCT of Personalized Fibre Diet in IBD
Brief Title: Personalized B-fructan Diet in Inflammatory Bowel Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B2022:074
Record Dates: First submitted 2022-10-04; First posted 2022-11-14 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Randomized pectin diet (Placebo Comparator)
  Interventions: Other: Placebo Comparator: Randomized pectin diet
- Randomized B-fructan diet (Placebo Comparator)
  Interventions: Other: Randomized B-fructan diet
- Personalized pectin diet (Experimental)
  Interventions: Other: Personalized pectin diet
- Personalized B-fructan diet (Experimental)
  Interventions: Other: Personalized B-fructan diet

INTERVENTIONS:
Other: Placebo Comparator: Randomized pectin diet — UC and healthy control participants randomized to receive recommendations provided by a dietician increasing consumption of foods high in pectin
  Arms: Randomized pectin diet
Other: Randomized B-fructan diet — UC and healthy control participants randomized to receive recommendations provided by a dietician increasing consumption of foods high in B-fructan
  Arms: Randomized B-fructan diet
Other: Personalized pectin diet — UC and healthy control participants to receive recommendations provided by a dietician increasing consumption of foods high in pectin based on personal host (biopsy) and microbe (stool) response at baseline
  Arms: Personalized pectin diet
Other: Personalized B-fructan diet — UC and healthy control participants to receive recommendations provided by a dietician increasing consumption of foods high in B-fructan based on personal host (biopsy) and microbe (stool) response at baseline
  Arms: Personalized B-fructan diet

SUMMARY:
This study aims to examine patient tolerability of personalized dietary fibre consumption recommendations (high-pectin diet versus high-B-fructan diet based on personalized responses), provided by an IBD dietician, based on our novel translational research findings.

ELIGIBILITY:
Inclusion Criteria:

* Children (age 6-17) or young adults (age 18-39).
* Known or suspected UC or IBDU [there will be 2 control group: non-IBD (undergoing colonoscopy but found not to have IBD; and healthy (no GI symptoms, so not required to have colonoscopy; could be family members)]
* For UC: Remission-mild-moderate disease: Mayo score <10
* Clinical indication for sedated colonoscopy
* Disease location: E2-E4
* Stable treatment (not on steroids; biologics or immunomodulator not changed in last month)
* High likelihood that patients will be able to collect all samples and provide all data

Exclusion Criteria:

* Use of antibiotics for a week or more over the last 3 months
* Use of probiotics or prebiotics at pharmacological doses (adding fibre sources to food or probiotics in yogurt, for example, are allowed)
* History of abdominal surgery, including appendectomy
* Documented enteric infection during the 3 months prior to endoscopy
* Presence of non-IBD bowel conditions (e.g., celiac), anatomical or mucosal abnormalities, motility disorder
* Presence of a systemic disease requiring treatment (cancer, ischemic heart disease, kidney failure, etc)
* Proctitis (E1)
* Systemic steroids (above 10 mg/day of Prednisone)
* Topical therapy within 1 week of endoscopy
* Recent change in IBD treatment (started biologics or IM over the last month)
* Pregnancy or planning to become pregnant during the study
* Inability to understand or sign the consent

Ages: 6 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Diet tolerability | 4 weeks
  Percentage of patients able to tolerate a personalized fiber diet provided by a dietitian will be evaluated at week 4 by measure of patient symptom score (PROMIS questionnaire) and willingness to continue adherence to diet advice provided.

SECONDARY OUTCOMES:
Inflammatory response to diet | 1 week, 4 weeks, 8 weeks, 12 weeks
  Host inflammatory response to personalized dietary fibre recommendations provided by dietitian will be determined by examining changes in markers of inflammation in blood and stool
Microbiota changes in response to diet | 1 week, 4 weeks, 8 weeks, 12 weeks
  Host microbiota response to personalized dietary fibre recommendations provided by dietitian will be determined by examining changes in microbe abundance, diversity and functions by shotgun metagenomics in stool

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Health Sciences Centre Hospital, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: Undecided